CLINICAL TRIAL: NCT06522087
Title: The Effect of 40 Hz Transcranial Stimulation on the Incidence of Delirium After Total Hip Replacement or Total Knee Replacement Arthroplasty in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Henan BJ
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Delirium; Anesthesia; Elderly
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40Hz stimulation group (Experimental): At the start of anesthesia, the subject received 40Hz transcranial stimulation for 1h.
  Interventions: Device: 40Hz stimulation
- Control group (No Intervention): At the start of anesthesia, the subject did not receive any additional treatment.

INTERVENTIONS:
Device: 40Hz stimulation — Exogenous 40HZ stimulation is a physical intervention that can drive oscillations in the gamma range, and the oscillations and pulses caused at the corresponding frequency can lead to a significant reduction in β-amyloid, reverse tau hyperphosphorylation, and thereby improve the cognitive function of patients.
  Arms: 40Hz stimulation group

SUMMARY:
Delirium is an acute confusional state, it is a sign of acute encephalopathy, also known as acute brain failure, acute brain dysfunction or mental state changes.Postoperative delirium can cause post-traumatic stress disorder, affects patients' quality of life, extend the length of hospital stay, increased hospitalization cost, and is closely relative to short-term and long-term mortality after surgery. Exogenous 40 Hz stimulation can improve cognitive functioning. Therefore, the aim of this study was to investigate the effect of exogenous 40Hz stimulation on the incidence of postoperative delirium in elderly patients undergoing hip and knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1.65-85 years old, gender not limited 2.General anesthesia unilateral total hip replacement surgery or unilateral total knee replacement 3.ASA classification I-III 4.No drugs for mental and central nervous system diseases were used before surgery 5.Preoperative MMSE score illiterate > 17 points, primary > 20 points, junior high school and above > 24 points 6.Obtaining informed consent

Exclusion Criteria:

1. Severe liver and kidney dysfunction
2. here were mental and nervous system diseases before operation
3. Have a history of alcoholism, long-term use of sedative or analgesic
4. A history of a delirium and other reasons are reluctant to cooperate
5. Massive blood loss and blood transfusion during operation, prolonged operation time

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Day 1, Day 2, Day 3 after surgery
  Postoperative delirium was assessed by CAM scale.The diagnosis of delirium mainly depends on four characteristics: 1 acute fluctuating course; 2 attention disorder; 3 thinking disorder; 4 change of consciousness level. At the same time, 1 and 2, and 3 or 4 can be used to diagnose delirium.

SECONDARY OUTCOMES:
Blood Markers | Preoperative and postoperative 1 d and 2 d
  Serum Tau proteomic analysis and CRP, IL-6, and B cell levels were recorded
The incidence of postoperative nausea and vomiting | Day 1, Day 2, Day 3 after surgery
  Follow up patients for nausea and vomiting
Sleep quality | Day 1, day 2, day 3 after surgery
  Sleep quality was assessed using a sleep quality scale(QS),(0: no effect on sleep 1: sleep in and out of sleep at night 2: sleep in and out of sleep unable to fall asleep 3: light sleep but unable to fall asleep 4: unable to fall asleep at all)
The incidence of pain | Day 1, day 2, day 3 after surgery
  NRS is a dotted ruler from 0 to 10. 0 means no pain, and 10 means unbearable pain. The patient chooses a number from above to describe the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan People's Hospital, Zhengzhou, Henan, China